CLINICAL TRIAL: NCT03359265
Title: Evaluate the Clinical Efficacy of Precious Metal Fiber Textile (Germanium Titanium π Element) for Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Juin-Hong Cherng, Assistant Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GREEN888
Record Dates: First submitted 2017-11-17; First posted 2017-12-02 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Active Comparator): The test group used underpants made of precious metal fibers (germanium, titanium and phosphorus), developed by Green Energy Nano Technology Co., Ltd.
  Interventions: Device: underpants
- Control (Placebo Comparator): The control group used commercially available underpants.
  Interventions: Device: underpants

INTERVENTIONS:
Device: underpants

SUMMARY:
Erectile dysfunction (ED) is common, and is defined as "persistent or regular inability to achieve or maintain penis erection for satisfactory intercourse". Approximately 3% to 71% of males have this problem as they age, and it is predicted that 320 million males worldwide will have ED by 2025. However, sex remains a topic that is too sensitive for most people to discuss openly. ED therapies include oral medication, vacuum erection devices, intracavernosal injection, testosterone supplementation, surgery, and psychological counseling. In addition, germanium (Ge), titanium (Ti), and π elements are noble metals that can be used to produce far-infrared radiation. There has been little application of these metals to the treatment of ED, but their use is worth investigating. Administered as health textiles, the application of these metals are expected to promote blood circulation, especially in the reproductive system, resulting in an improved sexual performance. Hence, the researcher aimed to investigate the safety and efficacy of Ge-Ti-π elements fiber textiles as an ED treatment, assessed by using the questionnaires related to the quality of sexual function.

DETAILED DESCRIPTION:
This clinical trial recruited 30 subjects with ED (a test group of 21 subjects and a control group of 9 subjects). Cellulosic textiles, incorporating noble metals (Ge, Ti, and π elements), developed by Green Energy Nano Technology Co., Ltd, were used in the test group, while commercially available regular textiles were used in the control group. The safety and efficacy of the treatment to the subject's sexual function quality were assessed through the International Index of Erectile Function (IIEF-5) and the validated Portuguese version of the Quality of Erection Questionnaire (QEQ) questionnaires. In the same session, the symptoms related to ED were assessed through the Premature Ejaculation Diagnostic Tool (PEDT) and the International Prostate Symptom Score (IPSS) questionnaires. The questionnaires were completed once a month and followed up for 3 months. The incidence of severe adverse effects was analyzed to assess product safety.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legal representative has understood the contents of this experiment and has agreed to sign the participation consent form.
2. The subject is aged between 40 and 70 years.
3. The patient has a medical history of erectile dysfunction for at least three months, based on a physician's diagnosis.
4. The subject has a regular sex partner during the experimental period.

Exclusion Criteria:

1. Subject was administered oral medication (Sildenafil, Vardenafil, or Tadalafil), vacuum suction device, or corpus cavernosum injections, seven days before the experiment commenced.
2. Long-term use of antihypertensive medication (doxazosin or nitrate), antidepressants, sedatives, anti-androgens, or medications such as cimetidine for digestive ulcers.
3. Severe damage to the central nervous system (including stroke or spinal injury) within the last six months.
4. Patients with erectile dysfunction induced by non-vascular causes, such as neurological factors, hormonal factors, or related trauma.
5. Patients with vascular sclerosis.
6. Patients with psychogenic erectile dysfunction.
7. Patients who had undergone radical prostatectomy or transurethral resection of the prostate.
8. HIV patients or patients with severe liver dysfunction (GOT, GPT ≥100 IU/L).
9. Patients with genital malformations or diseases that require sexual abstinence.
10. Sex partner is pregnant or nursing.
11. Patients with Peyronie's Disease.
12. Heavy drinkers or smokers.
13. Patients with malignant tumors or prostate cancer.
14. Patients who had surgery during the study period that could affect the experimental results.
15. Subjects who had a serious clinical or mental condition that could affect the experimental procedure or evaluation.

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 30 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The International Index of Erectile Function (IIEF-5) | 3 months
  IIEF-5 is a multidimensional validated questionnaire with 15 questions in the five domains of sexual function, such as erectile and orgasmic functions, sexual desire, satisfaction with intercourse, and overall sexual satisfaction. IIEF-5 scoring:
  The IIEF-5 score is the sum of the ordinal responses to the 5 items. 22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction
Quality of Erection Questionnaire (QEQ) | 3 months
  QEQ is a questionnaire that provides a further level of information by assessing satisfaction with the quality of the erections that were attained and maintained. QEQ is to be evaluated as a total score, which is the sum of responses to all items transformed onto a 5-30 scale.
  The maximum score on the QEQ is 30, and a higher score indicates better function.
Premature Ejaculation Diagnostic Tool (PEDT) | 3 months
  PEDT has been shown to be valid in detecting the presence of premature ejaculation among patients with five questions. Each item has a score of zero to four, and PEDT is scored by considering all five items together, which a higher score indicates highly suggestive of premature ejaculation.
International Prostate Symptom Score (IPSS) | 3 months
  IPSS is a well-known questionnaire to evaluate the symptom of prostate disease in patients. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).

CONTACTS AND LOCATIONS:
Locations (1):
- National Defense of Medical Center, Tri-Service General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Puppo V, Puppo G. Re: K. Hatzimouratidis, I. Eardley, F. Giuliano, et al. Guidelines on Male Sexual Dysfunction: Erectile Dysfunction and Premature Ejaculation. The Netherlands: European Association of Urology; 2015. http://uroweb.org/guideline/male-sexual-dysfunction/. Eur Urol. 2015 Dec;68(6):e136-7. doi: 10.1016/j.eururo.2015.08.026. Epub 2015 Aug 28. No abstract available. PMID 26320382
- [Background] Selvin E, Burnett AL, Platz EA. Prevalence and risk factors for erectile dysfunction in the US. Am J Med. 2007 Feb;120(2):151-7. doi: 10.1016/j.amjmed.2006.06.010. PMID 17275456
- [Background] Lewis RW. Epidemiology of sexual dysfunction in Asia compared to the rest of the world. Asian J Androl. 2011 Jan;13(1):152-8. doi: 10.1038/aja.2010.108. Epub 2010 Nov 15. PMID 21076440
- [Background] McKinlay JB. The worldwide prevalence and epidemiology of erectile dysfunction. Int J Impot Res. 2000 Oct;12 Suppl 4:S6-S11. doi: 10.1038/sj.ijir.3900567. PMID 11035380